CLINICAL TRIAL: NCT04393480
Title: Comparison of Upper Extremity Robotic Rehabilitation Efficiency With Conventional Rehabilitation in Patients With Hemiplegia After Cerebrovascular Event
Brief Title: Upper Extremity Robotic Rehabilitation in Patients With Hemiplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahel Taravati, M.D. (Other)
Responsible Party: Sponsor-Investigator, Sahel Taravati, M.D., Principal Investigator, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STKC2019
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Hemiplegia and/or Hemiparesis Following Stroke
Keywords: robotic therapy; rehabilitation; upper extremity; cerebrovascular event; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic therapy (Active Comparator): Robotic rehabilitation and conventional rehabilitation
  Interventions: Other: Robotic therapy; Other: Conventional therapy
- Conventional therapy (Sham Comparator): Conventional rehabilitation
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Robotic therapy — ReoGo™ - Motorika robotic therapy - upper extremity robotic rehabilitation system
  Arms: Robotic therapy
Other: Conventional therapy — Range of Motion (ROM) exercises, muscle strengthening, balance and mobility training, exercises for enhancing activities of daily life, neurophysiological exercises, turnings, bed movements, bridge building, sitting and transfer training, gait training, proprioceptive exercises, balance exercises on the balance board of those affected by the cerebellar system, occupational therapy, cognitive rehabilitation by the relevant psychologist given to those with cognitive impairment

SUMMARY:
Comparison of Upper Extremity Robotic Rehabilitation Efficiency with Conventional Rehabilitation in Patients with Hemiplegia after Cerebrovascular Event

DETAILED DESCRIPTION:
The aim of this single-blind randomized prospective study is to find out whether including robotic therapy in addition to conventional rehabilitation program has an effect on quality of life, motor function and activities of daily living of the hemiplegic patients. Hemiplegic patients diagnosed by anamnesis, physical examination and radiological analysis, which have been referred to the outpatient clinic of Ege University Faculty of Medicine Department of Physical Therapy and Rehabilitation between April 2016 and April 2019 have been taken to the study. The demographic and clinical data of the patients were recorded and they were randomized into 2 groups. 17 patients assigned to the robotic rehabilitation group (Study group) receiving robot-assisted rehabilitation in addition to conventional treatment and 20 assigned to the conventional rehabilitation group (control group) receiving only conventional therapy completed the study. Robotic-based rehabilitation given additionally was arranged to be 30-45 minutes, 5 days per week for 4 weeks. All patients were assessed at the beginning of therapy and at the end of 4th week with Brunnstrom stages of motor recovery, Fugl Meyer Assessment (FMA), hand grip strength, Purdue peg test, Minnesota manual dexterity test, Modified Ashworth Scale (MAS) , Functional Independance Measure (FIM), Stroke Specific Quality of Life Scale (SS-QOL), Nottingham Extended Activities of Daily Living (NEADL) Scale, Montreal Cognitive Assessment (MoCA), Center for Epidemiological Studies Depression Scale (CES- D). In the study, improvements in motor function scores, spasticity, general functioning, activities of daily living, cognitive assessment scale are better in robotic group when compared with control group but this difference was not statistically significant (p>0,05). The investigators have found statistically significant improvement in CES- Depression scale in robotic group compared with control group (p=0,018). Significantly improved motor function gains are observed before and after the treatment in both groups being better in the robotic group however no significant differences were observed between the groups after the treatment. Robotic rehabilitation provides a favorable alternative bringing slight benefits, and also advantageous in terms of work power and psychological recovery so robotic rehabilitation addition to conventional neurological rehabilitation is effective and useful in patient management after stroke or cerebrovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Having a single stroke
* Being an adult
* Having a duration of 4 to 30 months after stroke
* A score greater than 16 in mini-mental test
* Upper extremity Brunnstrom stage 2 or higher
* Being a fluent speaker in Turkish.

Exclusion Criteria:

* Severe apraxia
* Skin ulcers
* Multiple cerebrovascular events
* Severe decompensated diseases (cardiopulmonary, neurological, orthopedic and psychiatric etc), cardiac pacemakers, severe neuropsychological impairment,
* Neglect syndrome
* Spasticity greater than 3 in Modified Ashworth Scale
* Severe joint contractures
* Botulinum toxin-A injection in their upper extremity and dose change in drugs for spasticity in the last 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline hand grip strength at 4th week. | Up to 4 weeks
  Hand grip strength was measured using a hand dynamometer device(Jamar® Hand Dynamometer - Hydraulic - 200 lb Capacity). The measurements were recorded in kilograms. The higher scores indicates better outcome in hand grip strength.
Change from baseline hand functions (Minnesota manuel dexterity test) at 4th week. | Up to 4 weeks
  Manual Dexterity Test is a widely used test which measures the capacity for simple but rapid eye-hand-finger movement. This test includes two parts. The 'placing test' requires the patients to place 58 discs with a diameter of 3.5 cm in the spaces of another set of the same dimensions .The length of the sets requires a wide range of shoulder movements.The 'hand turning test' requires the patient to remove the discs from one set and place them in another, or to reinsert them by removing and turning them. This test was performed for the affected (hemiplegic side) upper limb of the patient (right or left) and the result was recorded in 'seconds'. Short periods show that the result is better.
Change from baseline hand functions (Purdue peg board) at 4th week. | Up to 4 weeks
  The Purdue Pegboard Test is a neuropsychological test of manual dexterity and bimanual coordination. The test involves two different abilities: gross movements of arms, hands, and fingers, and fine motor extremity. This test consists of a board with holes and pins that can be placed on them , also washers and nuts that can be attached to the pins. The patient is asked to insert as many pins as possible into the holes in 30 seconds in a straight row using his right hand.The same is then repeated for the left hand. Finally, by giving 1 minute time, it is passed to the stage where the patient inserts pins, nuts and washers by using two hands.The total score of these 3 stages gives the test score. The higher scores in this test shows better results.
Change from baseline spasticity (Modified Ashworth Scale (MAS)) at 4th week. | Up to 4 weeks
  The Modified Ashworth Scale is the most universally accepted clinical tool used to measure the increase of muscle tone. This scale is a numerical scale that grades spasticity from 0-4, with 0 being no resistance and 4 being a limb rigid in flexion or extension. The greater scores show increased spasticity and worse results.
Change from baseline neurophysiological development (Brunnstrom stage) at 4th week. | Up to 4 weeks
  The Brunnstrom Approach sets out a sequence of stages of recovery from hemiplegia after a stroke, emphasising the synergic pattern of movement which develops during recovery. It consists of six stages assessed separately for the upper limb, hand and lower limb. The higher scores show recovery and better results.
Change from baseline motor function (Fugl Meyer Assessment (FMA)) at 4th week. | Up to 4 weeks
  Fugl-Meyer Assessment (FMA) scale is an index to assess the sensorimotor impairment in individuals who have had stroke. The FMA motor assessments for the upper extremity consists of four subsections ( upper extremity, hand wrist, hand, speed/coordination). The total score ranges from 0 to 66, higher scores showing better motor function.
Change from baseline general function (Functional Independance Measure (FIM)) at 4th week. | Up to 4 weeks
  The Functional Independence Measure (FIM) is an 18-item measurement tool that explores an individual's physical, psychological and social function. Tasks that are evaluated using the FIM include six self-care activities, bowel and bladder control, transfers, locomotion, communication and social cognition. It is used to assess and grade the functional status of a person based on the level of assistance he or she requires. Grading categories range from "total assistance with helper"(score 0) to "complete independence with no helper"(score 7). The total score that can be obtained from this scale varies between 18-126, higher scores showing better results.
Change from baseline quality of life (Stroke Specific Quality of Life Scale (SS-QOL)) at 4th week. | Up to 4 weeks
  The Stroke Specific Quality Of Life scale (SS-QOL) is a patient-centered outcome measure intended to provide an assessment of health-related quality of life (HRQOL) specific to patients with stroke. SS-QOL contains 49 items and 12 fields; mobility, energy, upper limb function, work / production, mental state, self-care, social roles, family roles, vision, language, thinking and personality. Each field consists of at least 3 items, and each item is evaluated on a 5-point Likert scale. Higher scores reflect better function. The total score that can be obtained from SS-QOL varies between 49-245.
Change from baseline quality of life (Nottingham Extended Activities of Daily Living (NEADL)) at 4th week. | Up to 4 weeks
  The Nottingham Extended Activities of Daily Living (NEADL scale) comprises 22 questions to measure the independence in the following areas of daily living: mobility, kitchen, domestic and leisure activities. The total score varies between 0-66. Higher scores show better outcome.
Change from baseline cognitive state (MoCA test) at 4th week. | Up to 4 weeks
  The Montreal Cognitive Assessment (MoCA) is a brief 30-question test that takes around 10 to 12 minutes to complete and helps assess people for cognitive impairment. Different cognitive functions are evaluated with MoCA. These are attention, memory, concentration, executive functions, language functions, visual structuring skills, abstract thinking, computation and orientation. The score varies between 0 and 30 points and patients who get 21 points and above are considered normal. Higher scores indicate better results.
Change from baseline emotional state (CES-depression test) at 4th week. | Up to 4 weeks
  CES-depression test is a quick self-test, consisting of 20 items that measure depressive feelings and behaviours during the past week and one of the most common screening tests for helping an individual to determine his or her depression quotient.
  With the four-dimensional structure of the scale, depressive symptoms, positive effects, somatic symptoms and difficulties in interpersonal relationships were aimed to be measured. Score ranges from 0 to 60, and high scores indicate depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahel Taravati, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Özcan O, Arpacıoğlu O, et al. Nörorehabilitasyon: Güneş & Nobel Tıp Kitabevleri; 2000
- [Background] Oğuz H, Dursun E, et al. Tıbbi rehabilitasyon: Nobel Tıp Kitabevleri; 2004
- [Background] Norouzi-Gheidari N, Archambault PS, Fung J. Effects of robot-assisted therapy on stroke rehabilitation in upper limbs: systematic review and meta-analysis of the literature. J Rehabil Res Dev. 2012;49(4):479-96. doi: 10.1682/jrrd.2010.10.0210. PMID 22773253
- [Background] Rosati G, Oscari F, Reinkensmeyer DJ, Secoli R, Avanzini F, Spagnol S, Masiero S. Improving robotics for neurorehabilitation: enhancing engagement, performance, and learning with auditory feedback. IEEE Int Conf Rehabil Robot. 2011;2011:5975373. doi: 10.1109/ICORR.2011.5975373. PMID 22275577
- [Background] Aisen ML, Krebs HI, Hogan N, McDowell F, Volpe BT. The effect of robot-assisted therapy and rehabilitative training on motor recovery following stroke. Arch Neurol. 1997 Apr;54(4):443-6. doi: 10.1001/archneur.1997.00550160075019. PMID 9109746
- [Background] Lo AC, Guarino PD, Richards LG, Haselkorn JK, Wittenberg GF, Federman DG, Ringer RJ, Wagner TH, Krebs HI, Volpe BT, Bever CT Jr, Bravata DM, Duncan PW, Corn BH, Maffucci AD, Nadeau SE, Conroy SS, Powell JM, Huang GD, Peduzzi P. Robot-assisted therapy for long-term upper-limb impairment after stroke. N Engl J Med. 2010 May 13;362(19):1772-83. doi: 10.1056/NEJMoa0911341. Epub 2010 Apr 16. PMID 20400552
- [Background] Nef T., Klamroth-Marganska V., Keller U., Riener R. (2016) Three-Dimensional Multi-degree-of-Freedom Arm Therapy Robot (ARMin). In: Reinkensmeyer D., Dietz V. (eds) Neurorehabilitation Technology. Springer, Cham
- [Background] Chang WH, Kim YH. Robot-assisted Therapy in Stroke Rehabilitation. J Stroke. 2013 Sep;15(3):174-81. doi: 10.5853/jos.2013.15.3.174. Epub 2013 Sep 27. PMID 24396811
- [Background] Teasell R, Foley N, Salter K, Bhogal S, Jutai J, Speechley M. Evidence-Based Review of Stroke Rehabilitation: executive summary, 12th edition. Top Stroke Rehabil. 2009 Nov-Dec;16(6):463-88. doi: 10.1310/tsr1606-463. No abstract available. PMID 20139049
- [Background] Lum PS, Burgar CG, Shor PC, Majmundar M, Van der Loos M. Robot-assisted movement training compared with conventional therapy techniques for the rehabilitation of upper-limb motor function after stroke. Arch Phys Med Rehabil. 2002 Jul;83(7):952-9. doi: 10.1053/apmr.2001.33101. PMID 12098155
- [Background] Teasell R, Bayona N, et al. Background concepts in stroke rehabilitation. Evidence-Based Review of Stroke Rehabilitation. 2008
- [Background] Masiero S, Armani M, Ferlini G, Rosati G, Rossi A. Randomized trial of a robotic assistive device for the upper extremity during early inpatient stroke rehabilitation. Neurorehabil Neural Repair. 2014 May;28(4):377-86. doi: 10.1177/1545968313513073. Epub 2013 Dec 6. PMID 24316679
- [Background] Taveggia G, Borboni A, Salvi L, Mule C, Fogliaresi S, Villafane JH, Casale R. Efficacy of robot-assisted rehabilitation for the functional recovery of the upper limb in post-stroke patients: a randomized controlled study. Eur J Phys Rehabil Med. 2016 Dec;52(6):767-773. Epub 2016 Jul 13. PMID 27406879
- [Background] Veerbeek JM, Langbroek-Amersfoort AC, van Wegen EE, Meskers CG, Kwakkel G. Effects of Robot-Assisted Therapy for the Upper Limb After Stroke. Neurorehabil Neural Repair. 2017 Feb;31(2):107-121. doi: 10.1177/1545968316666957. Epub 2016 Sep 24. PMID 27597165
- [Background] Prange GB, Jannink MJ, Groothuis-Oudshoorn CG, Hermens HJ, Ijzerman MJ. Systematic review of the effect of robot-aided therapy on recovery of the hemiparetic arm after stroke. J Rehabil Res Dev. 2006 Mar-Apr;43(2):171-84. doi: 10.1682/jrrd.2005.04.0076. PMID 16847784
- [Background] Bertani R, Melegari C, De Cola MC, Bramanti A, Bramanti P, Calabro RS. Effects of robot-assisted upper limb rehabilitation in stroke patients: a systematic review with meta-analysis. Neurol Sci. 2017 Sep;38(9):1561-1569. doi: 10.1007/s10072-017-2995-5. Epub 2017 May 24. PMID 28540536
- [Background] Poli P, Morone G, Rosati G, Masiero S. Robotic technologies and rehabilitation: new tools for stroke patients' therapy. Biomed Res Int. 2013;2013:153872. doi: 10.1155/2013/153872. Epub 2013 Nov 20. PMID 24350244
- [Background] Klamroth-Marganska V, Blanco J, Campen K, Curt A, Dietz V, Ettlin T, Felder M, Fellinghauer B, Guidali M, Kollmar A, Luft A, Nef T, Schuster-Amft C, Stahel W, Riener R. Three-dimensional, task-specific robot therapy of the arm after stroke: a multicentre, parallel-group randomised trial. Lancet Neurol. 2014 Feb;13(2):159-66. doi: 10.1016/S1474-4422(13)70305-3. Epub 2013 Dec 30. PMID 24382580
- [Background] Takahashi K, Domen K, Sakamoto T, Toshima M, Otaka Y, Seto M, Irie K, Haga B, Takebayashi T, Hachisuka K. Efficacy of Upper Extremity Robotic Therapy in Subacute Poststroke Hemiplegia: An Exploratory Randomized Trial. Stroke. 2016 May;47(5):1385-8. doi: 10.1161/STROKEAHA.115.012520. Epub 2016 Mar 22. PMID 27006452
- [Background] Tomic TJ, Savic AM, Vidakovic AS, Rodic SZ, Isakovic MS, Rodriguez-de-Pablo C, Keller T, Konstantinovic LM. ArmAssist Robotic System versus Matched Conventional Therapy for Poststroke Upper Limb Rehabilitation: A Randomized Clinical Trial. Biomed Res Int. 2017;2017:7659893. doi: 10.1155/2017/7659893. Epub 2017 Jan 31. PMID 28251157
- [Background] Zhang C, Li-Tsang CW, Au RK. Robotic approaches for the rehabilitation of upper limb recovery after stroke: a systematic review and meta-analysis. Int J Rehabil Res. 2017 Mar;40(1):19-28. doi: 10.1097/MRR.0000000000000204. PMID 27926617
- [Background] Kwakkel G, Kollen BJ, Krebs HI. Effects of robot-assisted therapy on upper limb recovery after stroke: a systematic review. Neurorehabil Neural Repair. 2008 Mar-Apr;22(2):111-21. doi: 10.1177/1545968307305457. Epub 2007 Sep 17. PMID 17876068
- [Derived] Taravati S, Capaci K, Uzumcugil H, Tanigor G. Evaluation of an upper limb robotic rehabilitation program on motor functions, quality of life, cognition, and emotional status in patients with stroke: a randomized controlled study. Neurol Sci. 2022 Feb;43(2):1177-1188. doi: 10.1007/s10072-021-05431-8. Epub 2021 Jul 11. PMID 34247295